CLINICAL TRIAL: NCT03454802
Title: Passive Leg Raising - an Important Diagnostic Manoeuvre and Its Dependency on the Activity of the Autonomous Nervous System in Critically Ill Patients and Healthy Subjects
Brief Title: Passive Leg Raising - an Important Diagnostic Manoeuvre
Acronym: PLR-ANS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Region MidtJylland Denmark (Other)
Collaborators: Edwards Lifesciences (Industry)
Responsible Party: Principal Investigator, Soren Sondergaard, Senior Consultant, MD, PhD, Region MidtJylland Denmark
Allocation: Non-Randomized | Model: Sequential | Masking: Single | Purpose: Basic Science
Other Study IDs: 619909
Record Dates: First submitted 2018-02-10; First posted 2018-03-06 (Actual); Last update posted 2021-09-24 (Actual); Status verified 2021-09

CONDITIONS: Cardiovascular Insufficiency

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (3):
- Normal subjects (Active Comparator): Normal subjects 'Passive Leg Raising'
  Interventions: Diagnostic Test: Passive Leg Raising
- ICU patients (Active Comparator): ICU patients 'Passive Leg Raising'
  Interventions: Diagnostic Test: Passive Leg Raising
- Cardiac Outpatients (Active Comparator): Cardiac Outpatients 'Passive Leg Raising'
  Interventions: Diagnostic Test: Passive Leg Raising

INTERVENTIONS:
Diagnostic Test: Passive Leg Raising — See above

SUMMARY:
The aim is to describe the physiological background for PLR and the interpretation of a PLR manoeuvre.

The protocol entails the measurement of stroke volume (SV) at baseline (semirecumbent patient position), during PLR and after returning to semirecumbent position. Simultaneously blood pressure (BP), pulse rate (PR), pulse oximetric saturation (SpO2) and ECG are recorded. The procedure is performed in ten normal subjects, ten patients recruited in the cardiology outpatient department and ten critically ill patients under analgosedation in the ICU.

Analysis includes changes in measured variables and heart rate variability in the frequency domain during the three phases of the experiment.

DETAILED DESCRIPTION:
See above

ELIGIBILITY:
Inclusion Criteria:

Consenting after written and oral information

Exclusion Criteria:

Contraindications to PLR: intracranial or abdominal hypertension

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2020-10-01 (Actual); Study Completion 2020-10-01 (Actual)

PRIMARY OUTCOMES:
Changes in cardiovascular variables I | 10 minutes
  stroke volume, SV (mL)
Changes in cardiovascular variables II | 10 minutes
  pulse rate, PR (min^-1)
Changes in cardiovascular variables III | 10 minutes
  blood pressure, BP (mmHg)
Changes in cardiovascular variables IV | 10 minutes
  pulse oximetric saturation, SpO2 (%)
Changes in HRV frequency domain variables V | 10 minutes
  Heart rate variability, HRV, variables in frequency domain (low frequency, LF, 0.04-0.15 Hz, high frequency, HF, 0.15-0.4 Hz)
Changes in HRV frequency domain variables VI | 10 minutes
  HRV absolute power (ms^2, natural logarithm transformed values of absolute powers of very low frequency, VLF, LF, and HF bands)
Changes in HRV frequency domain variables VII | 10 minutes
  HRV relative power (absolute power/total power)
Changes in HRV frequency domain variables VIII | 10 minutes
  HRV normalized power (%, normalized units, n.u.)
Changes in HRV frequency domain variables IX | 10 minutes
  HRV total power given by VLF + HF + LF (ms2) and LF/HF ratio.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Toft, MD, Study Chair — Head of Centre of Planned Surgery, Silkeborg Regional Hospital
Locations (1):
- Regionshospitalet Silkeborg, Silkeborg, Central Jutland, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Monnet X, Rienzo M, Osman D, Anguel N, Richard C, Pinsky MR, Teboul JL. Passive leg raising predicts fluid responsiveness in the critically ill. Crit Care Med. 2006 May;34(5):1402-7. doi: 10.1097/01.CCM.0000215453.11735.06. PMID 16540963